CLINICAL TRIAL: NCT03817307
Title: Validation of USPIO-enhanced MRI for Detection of Lymph Node Metastases in Head and Neck Carcinoma: A Pilot Study
Brief Title: Validation of USPIO-enhanced MRI for Detection of Lymph Node Metastases in Head and Neck Carcinoma
Acronym: USPIO-NECK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USPIO-NECK
Record Dates: First submitted 2018-12-20; First posted 2019-01-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- USPIO enhanced-MRI (Experimental): The contrast agent ferumoxtran-10 will be administered intravenously under constant medical supervision 24-36 hours before performing a T2* weighted MRI scan (prior to surgery).
  Interventions: Diagnostic Test: USPIO-enhanced MRI

INTERVENTIONS:
Diagnostic Test: USPIO-enhanced MRI — The USPIO contrast agent will be administered intravenously to the subjects. An MRI scan of the neck region is performed 24-36 hours later to detect lymph node metastases.

SUMMARY:
This study evaluates the diagnostic accuracy of USPIO enhanced MRI for the detection of lymph node metastases in head-and-neck squamous cell carcinoma (SCC) using histopathology as a gold standard.

DETAILED DESCRIPTION:
The presence of lymph node metastases has a large impact on prognosis and treatment in head-and neck cancer patients and necessitates treatment intensification. Determining lymph node status, however, is a challenge because up to 20% of patients with a pre-operative clinically negative neck will have occult metastases in the neck dissection specimen. One promising technique is USPIO-enhanced MRI, an MR-imaging technique in which ultrasmall superparamagnetic iron oxide (USPIO) particles are intravenously infused as a contrast agent in patients 24-36 hours before the MRI examination and has proven to be of value in detecting lymph node metastases in various types of cancer. The investigators want to validate this technique in a cohort of head and neck cancer patients who undergo neck dissection surgery. Histopathology wills serve as the gold standard and the correlation will be made on a (neck)level-to-level and node-to-node basis. Since the investigators have no experience in reading USPIO-enhanced MR images of the neck with 3-dimensional iron-sensitive MR sequences, this study starts with an explorative part and will be followed by the pilot study. The explorative component aims at obtaining knowledge regarding visual features of (non-)metastatic cervical lymph nodes on USPIO-enhanced MR images. The purpose is that the observers work through a learning curve. The information obtained will be used to develop a scoring system for the radiologic assessment of cervical lymph nodes in the subsequent part of our study.

If USPIO-enhanced MRI is successful, this may obviate the need for a sentinel node procedure for example. Furthermore, it could guide treatment such as the performance of more selective neck dissections and de-escalation of the radiation dose to healthy tissues in order to decrease morbidity but maintaining high cure rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically proven cT0-4N0-3M0 SCC of the oral cavity, oropharynx, hypopharynx, larynx or unknown primary.
* Patients planned to undergo a neck dissection.
* Patient provided written informed consent.

Exclusion Criteria:

* Patients who underwent radio- and/or chemotherapy to the neck before surgery.
* Patients who had a previous lymphadenectomy in the head and neck region.
* Patients with contraindications to MRI (epilepsy; claustrophobia; metallic splinters; pacemaker, pacemaker wires or implanted defibrillator; implanted magnets in jaw; arterial clips (carotid arteries); pregnancy; auditory implant, neurogenic bladder stimulator, insulin pump, neurostimulator, baclofen pump; metallic tissue expander after mastectomy; cochlear implant; metallic braces; other foreign bodies implanted)
* Patients with contraindications to USPIO based contrast agents (prior allergic reaction to ferumoxtran-10 or any other iron preparation; prior allergic reaction attributed to dextran or other polysaccharide, in any preparation; hereditary hemochromatosis, hemosiderosis, chronic hemolytic anaemia (e.g. thalassemia, sickle cell anaemia); pregnancy)
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of USPIO-enhanced MRI for detecting lymph node metastases on a level basis. | The data of each patient will be assessed prior to neck dissection surgery.
  The images of the USPIO-enhanced MRI will be read by two radiologists who will score each level as cancer (metastases) positive or negative. These results will be compared with the results of pathology which serve as the gold standard to determine the sensitivity, specificity, positive predictive value and negative predictive value of the USPIO-enhanced MRI for detecting lymph node metastases in head-and-neck cancer patients.

SECONDARY OUTCOMES:
Diagnostic accuracy of USPIO-enhanced MRI for detecting lymph node metastases on a nodal basis. | The data of each patient will be assessed prior to neck dissection surgery.
  The images of the USPIO-enhanced MRI will be read by two radiologists who will score each node as cancer (metastases) positive or negative. These results will be compared with the results of pathology which serve as the gold standard to determine the sensitivity, specificity, positive predictive value and negative predictive value of the USPIO-enhanced MRI for detecting lymph node metastases in head-and-neck cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dijkema, MD, PhD, Principal Investigator — Radboud University Medical Center; Hans Kaanders, Prof, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Derived] Driessen DAJJ, Zamecnik P, Dijkema T, Pegge SAH, van Engen-van Grunsven ACH, Takes RP, Kaanders JHAM, Scheenen TWJ. High-Accuracy Nodal Staging of Head and Neck Cancer With USPIO-Enhanced MRI: A New Reading Algorithm Based on Node-to-Node Matched Histopathology. Invest Radiol. 2022 Dec 1;57(12):810-818. doi: 10.1097/RLI.0000000000000902. Epub 2022 Jul 1. PMID 35776432